CLINICAL TRIAL: NCT01491191
Title: Perioperative Use of Palmitoylethanolamide for Prevention of Chronic Postsurgical Pain in Patients Undergoing Elective Surgery.
Brief Title: Palmitoylethanolamide for Post-operative Pain Prevention
Acronym: PEAforCPSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Laura Rinaldi, Medical Doctor, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 213/11
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Post-operative Pain
Keywords: surgical pain; chronic pain; prevention; palmitoylethanolamide
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — palmidrol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEA (Experimental): Administration of PEA from 8 days before surgical operation until 30 days after surgery.
  Interventions: Dietary Supplement: Palmitoylethanolamide
- Sugar pill (Active Comparator): Administration of placebo from 8 days before surgical operation until 30 days after surgery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Palmitoylethanolamide — Before surgery: 600 mg cp twice a day After surgery: 600 mg microgranules twice a day for 10 days then 600 mg cps once a day for 20 days
  Arms: PEA
Dietary Supplement: Placebo — Before surgery: 1 sugar pill twice a day for 8 days After surgery: 1 sugar microgranules twice a day for 10 days then 1 sugar pill once a day for 20 days
  Arms: Sugar pill

SUMMARY:
Postsurgical pain becomes chronic when it lasts more then two months after surgery. A neurogenic or neuropathic pathogenesis is hypothesized for this event that reaches high rates after urologic and gynecologic surgeries.

Palmitoylethanolamide (PEA) binds to mast cells and regulates pro-inflammatory factors release, without adverse events.

The investigators assume that perioperative administration of PEA can reduce chronic postsurgical pain incidence of patients undergoing to urologic and gynecologic elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective gynecological or urological surgical procedures

Exclusion Criteria:

* age < 18
* pregnancy or nursing
* pre-existing chronic pain
* severe hepatic or renal failure
* post-operative progression of local cancer disease
* post-operative infection or inflammation of surgical wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of chronic post-surgical pain | 2 months after surgery
  Assessment of pain persisting in surgical site after uncomplicated postoperative healing. Assessment of skin hyperalgesia about the surgical wound.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Rinaldi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Policlinico di Modena; Alberto Pasetto, PhD, Study Director — Azienda Ospedaliero-Universitaria Policlinico di Modena
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena, Modena, Italy